CLINICAL TRIAL: NCT06549816
Title: An Open-label, Phase 1 Study to Investigate the Safety and Pharmacokinetics of SGN-B6A in Chinese Subjects With Advanced Solid Tumors
Brief Title: A Study of SGN-B6A in Chinese Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGNB6A-003; C5751004 (Other: Alias Study Number)
Record Dates: First submitted 2024-07-22; First posted 2024-08-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Esophageal Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: NSCL; Lung Neoplasm; Cancer of Ovary; Ovarian Cancer; Colorectal Cancer; Colorectal Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus; Lung Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sigvotatug vedotin (Experimental): sigvotatug vedotin monotherapy 1.8 mg/kg adjusted ideal body weight intravenous administration on Days 1 and 15 of a 28-day cycle.
  Interventions: Drug: sigvotatug vedotin

INTERVENTIONS:
Drug: sigvotatug vedotin — Sigvotatug vedotin is a antibody-drug conjugate (ADC) designed to deliver the cytotoxic agent monomethyl auristatin E (MMAE) to cells expressing integrin beta-6.

SUMMARY:
This trial will look at a drug called sigvotatug vedotin (SGN-B6A) to find out whether it is safe for Chinese participants who have solid tumors. It will study sigvotatug vedotin to find out what its side effects are. A side effect is anything the drug does besides treating cancer. It will also study how do Chinese participants' body interact with sigvotatug vedotin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed metastatic or unresectable locally advanced solid malignancy within one of the tumor types listed below.

  * NSCLC
  * HNSCC
  * ESCC
  * GAC
  * EAC
  * GEJ adenocarcinoma
* Subjects must have disease that is relapsed or refractory, or be intolerant to systemic standard-of-care therapies, and in the judgement of the investigator, should have no appropriate standard-of-care therapeutic option. If a standard-of-care therapy is available that has not been administered, the reason that the therapy is not appropriate must be documented.
* Adequate organ function as defined by the baseline laboratory criteria obtained within 7 days prior to SGN-B6A initiation (Cycle 1 Day 1)
* Measurable or non-measurable disease per RECIST v1.1 at baseline.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.

Exclusion Criteria:

* History of another malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Participants with any of the following respiratory conditions:

  * Evidence of noninfectious interstitial lung disease (ILD) or pneumonitis that:
  * * Was previous diagnosed and required systemic steroids, or
  * * Is currently diagnosed and managed, or
  * * Is suspected on radiologic imaging at screening
  * Known diffusing capacity of the lung for carbon monoxide (DLCO) < 50%
  * Any Grade greater than or equal to (≥) 3 pulmonary disease unrelated to underlying malignancy
  * Prior radiation therapy to the lung that is >30 gray (Gy) within 6 months of the first dose of sigvotatug vedotin.
* Pre-existing peripheral neuropathy Grade greater than or equal to (≥) 2
* Uncontrolled diabetes mellitus
* Known active central nervous system metastases. Participants with previously treated brain metastases may participate provided they:

  * are clinically stable for at least 4 weeks prior to study entry after brain metastasis treatment,
  * have no new or enlarging brain metastases, and
  * are off of corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to first dose of study drug.
* Known history or current diagnosis of carcinomatous meningitis
* Previous treatment with an MMAE-containing agent or an agent targeting integrin beta-6
* Prior anticancer therapies:

  * Chemotherapy within 21 days prior to first administration of sigvotatug vedotin
  * Targeted small molecule agents within 14 days or 5 half-lives (whichever is longer) prior to first administration of sigvotatug vedotin
  * Antibody-based anticancer or other investigational antitumor therapy within 28 days prior to first administration of sigvotatug vedotin
  * Focal radiotherapy or major surgery that is not completed 14 days prior to the first dose of sigvotatug vedotin
* Traditional or herbal medicines:

  * Anti-cancer traditional or herbal medicines within 28 days prior to first administration of sigvotatug vedotin
  * Traditional or herbal medicines for other purposes (such as supportive care) within 7 days prior to first administration of sigvotatug vedotin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants with laboratory abnormalities | Through 30-37 days following last dose of sigvotatug vedotin; up to 3 years
Number of participants with dose-limiting toxicities (DLTs) | Up to 28 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of antibody-conjugated monomethyl auristatin E (ac-MMAE) in plasma: Area under the curve (AUC) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 through predose Cycle 1 Day 15; Multiple dose: Cycle 2 Day 1 through predose Cycle 2 Day 15 (Each Cycle is 28 days)
PK of ac-MMAE in plasma: maximum concentration (Cmax) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 (predose, end of infusion [EOI], and 2 hour and 4 hour post-dose); Multiple dose: Cycle 2 Day 1 (predose, EOI, and 2 hour and 4 hour post-dose) (Each Cycle is 28 days)
PK of ac-MMAE in plasma: time to maximum concentration (Tmax) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 (predose, End of Infusion (EOI), and 2 hour and 4 hour post-dose); Multiple dose: Cycle 2 Day 1 (predose, EOI, and 2 hour and 4 hour post-dose) (Each Cycle is 28 days)
PK of ac-MMAE in plasma: apparent half-life (t1/2) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 through predose Cycle 1 Day 15; Multiple dose: Cycle 2 Day 1 through predose Cycle 2 Day 15 (Each Cycle is 28 days)
PK of ac-MMAE in plasma: trough concentration (Ctrough) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 15 predose; Multiple dose: Cycle 2 Day 15 predose (Each Cycle is 28 days)
PK of monomethyl auristatin E (MMAE) in plasma - AUC after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 through predose Cycle 1 Day 15; Multiple dose: Cycle 2 Day 1 through predose Cycle 2 Day 15 (Each Cycle is 28 days)
PK of MMAE in plasma: maximum concentration (Cmax) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 (predose, end of infusion [EOI], and 2 hour and 4 hour post-dose); Multiple dose: Cycle 2 Day 1 (predose, EOI, and 2 hour and 4 hour post-dose) (Each Cycle is 28 days)
PK of MMAE in plasma: time to maximum concentration (Tmax) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 (predose, EOI, and 2 hour and 4 hour post-dose); Multiple dose: Cycle 2 Day 1 (predose, EOI, and 2 hour and 4 hour post-dose) (Each Cycle is 28 days)
PK of MMAE in plasma: apparent half-life (t1/2) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 1 through predose Cycle 1 Day 15; Multiple dose: Cycle 2 Day 1 through predose Cycle 2 Day 15 (Each Cycle is 28 days)
PK of MMAE in plasma: trough concentration (Ctrough) after a single dose and multiple doses of SGN-B6A | Single dose: Cycle 1 Day 15 predose; Multiple dose: Cycle 2 Day 15 predose (Each Cycle is 28 days)
Number of participants with antidrug antibodies | From first dose through up to 37 days following last dose of sigvotatug vedotin

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- China (3):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNB6A-003